CLINICAL TRIAL: NCT03019588
Title: A Phase III, Randomized, Open-label Clinical Trial of Pembrolizumab (MK-3475) Versus Paclitaxel in Asian Subjects With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Who Progressed After First-Line Therapy With Platinum and Fluoropyrimidine
Brief Title: Efficacy and Safety Study of Pembrolizumab (MK-3475) Versus Paclitaxel in Asian Participants With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma Who Progressed After First-line Therapy With Platinum and Fluoropyrimidine (MK-3475-063/KEYNOTE-063)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-063; MK-3475-063 (Other: Merck Protocol Number)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Results first posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2022-06

CONDITIONS: Gastric Neoplasms; Gastroesophageal Junction Adenocarcinoma
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Stomach Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab 200 mg (Experimental): Participants receive pembrolizumab 200 mg intravenous (IV) infusion on Day 1 of each 3-week cycle for up to 35 cycles (up to approximately 2 years).
  Interventions: Biological: Pembrolizumab
- Paclitaxel 80 mg/m^2 (Active Comparator): Participants receive paclitaxel 80 mg/m^2 IV infusion on Days 1, 8 and 15 of each 4-week cycle for up to approximately 2 years.
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475
  Arms: Pembrolizumab 200 mg
Drug: Paclitaxel — IV infusion
  Arms: Paclitaxel 80 mg/m^2

SUMMARY:
The study will compare the efficacy and safety of treatment with pembrolizumab (MK-3475) versus paclitaxel in Asian, programmed death-ligand 1 (PD-L1) positive participants with advanced gastric or gastroesophageal junction (GEJ) adenocarcinoma who have progressed after failure of any combination chemotherapy containing a platinum and a fluoropyrimidine agent.

The primary study hypotheses are that pembrolizumab prolongs Overall Survival (OS) compared to paclitaxel and that pembrolizumab prolongs Progression-free Survival (PFS) per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) assessed by blinded central radiologists' review compared to paclitaxel.

DETAILED DESCRIPTION:
Once the participant has achieved the study objective or the study has ended, the participant will be discontinued from the study and may be enrolled in an extension study to continue protocol-defined assessments and treatment. Enrollment in the extension study will be conditional on participant consent. Treatment with pembrolizumab or paclitaxel will continue until documented disease progression, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to discontinue the participant, participant withdraws consent, pregnancy of the participant, participant receives 35 administrations (approximately 2 years) of pembrolizumab, or administrative reasons requiring cessation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically-confirmed diagnosis of gastric or GEJ adenocarcinoma.
* Has metastatic disease or locally advanced, unresectable disease.
* Has measurable disease as defined by RECIST 1.1 as determined by investigator.
* Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale within 3 days prior to the first dose of study treatment.
* Has experienced documented objective radiographic or clinical disease progression during or after first-line therapy containing any platinum/fluoropyrimidine doublet.
* Is willing to provide tissue for PD-L1 biomarker analysis.
* Has PD-L1 positive tumor (based on analysis of sample provided to core lab).
* Female participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment for the pembrolizumab arm and through 180 days after the last dose of study treatment for the paclitaxel arm.
* Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study treatment for the pembrolizumab arm and through 180 days after the last dose of study treatment for the paclitaxel arm.
* Demonstrates adequate organ function.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of trial treatment.
* Has squamous cell or undifferentiated gastric cancer.
* Has active autoimmune disease that has required systemic treatment in past 2 years.
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤ Grade 1 or at Baseline) from AEs due to agents administered more than 4 weeks earlier.
* Has had prior chemotherapy, targeted small molecule therapy, radiation therapy, or any other agents used as systemic treatment for cancer, within 2 weeks prior to the first dose of trial treatment or who has not recovered (i.e., ≤ Grade 1 or at Baseline) from AEs due to a previously administered agent.
* Has a known additional malignancy that is progressing or has required active treatment within the past 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has an active infection requiring systemic therapy.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment for the pembrolizumab arm and through 180 days after the last dose of study treatment for the paclitaxel arm.
* Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g. cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137).
* Has a known history of Human Immunodeficiency Virus (HIV) infection.
* Has known active Hepatitis B or C virus infection.
* Has received a live vaccine within 30 days of planned start of study treatment.
* Has known allergy or hypersensitivity to paclitaxel or any components used in the paclitaxel preparation or other contraindication for taxane therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (36):
- China (25):
  - Beijing Cancer Hospital ( Site 0022), Beijing, Beijing Municipality
  - Fuzhou General Hospital of Nanjing Military Command ( Site 0023), Fuzhou, Fujian
  - The First People's Hospital of Changzhou ( Site 0024), Changzhou, Jiangsu
  - Nanjing 81 PLA Hospital, Dept. of Oncology ( Site 0001), Nanjing, Jiangsu
  - Jilin Province Cancer Hospital, Department of Chemotherapy ( Site 0002), Changchun, Jilin
  - Tangdu Hospital ( Site 0030), Xi’an, Shanxi
  - 2nd Affil Hosp of Zhejiang University College of Medicine ( Site 0014), Hangzhou, Zhejiang
  - 301 Hospital ( Site 0008), Beijing
  - 307 Hospital of PLA, Dept. of Oncology ( Site 0006), Beijing
  - Peking Union Medical College Hospital ( Site 0011), Beijing
  - Xiangya Hospital Central -South University ( Site 0021), Changsha
  - Sir Sun Sun Shaw Hosp, Zhejiang Univ,Oncology dept. ( Site 0016), Hangzhou
  - The First Affiliated Hospital of Zhejiang University ( Site 0004), Hangzhou
  - Harbin Medical University Cancer Hospital ( Site 0020), Harbin
  - Anhui Provincial Hospital ( Site 0017), Hefei
  - The First Affiliated Hospital of Anhui Medical University ( Site 0012), Hefei
  - The Second Hospital of Anhui Medical University ( Site 0013), Hefei
  - Jiangsu Cancer Hospital ( Site 0003), Nanjing
  - Renji Hospital Shanghai Jiaotong University School of Medicine ( Site 0028), Shanghai
  - Ruijin Hospital, Shanghai Jiaotong University ( Site 0018), Shanghai
  - Shanghai East Hospital ( Site 0033), Shanghai
  - Shanghai Tenth People's Hospital ( Site 0026), Shanghai
  - Zhongshan Hospital affiliated to Fudan University ( Site 0005), Shanghai
  - Shanghai First People's Hospital ( Site 0027), Songjiang
  - Tongji Medical College Huazhong Uinversity Of Science and Technology ( Site 0025), Wuhan
- University Malaya Medical Centre (UMMC) ( Site 0126), Kuala Lumpur, Kuala Lumpur, Malaysia
- South Korea (6):
  - National Cancer Center ( Site 0202), Goyang-si, Gyeonggi-do
  - CHA Bundang Medical Center CHA University ( Site 0203), Seongnam-si, Gyeonggi-do
  - The Catholic University of Korea, St. Vincent's Hospital ( Site 0201), Suwon, Gyeonggi-do
  - Asan Medical Center ( Site 0204), Seoul
  - Kangbuk Samsung Hospital ( Site 0205), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0206), Seoul
- Taiwan (4):
  - Chang Gung Medical Foundation - Kaohsiung ( Site 0227), Kaohsiung City
  - China Medical University Hospital. ( Site 0226), Taichung
  - Koo Foundation Sun Yat-Sen Cancer Center ( Site 0228), Taipei
  - MacKay Memorial Hospital ( Site 0229), Taipei

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Chung HC, Kang YK, Chen Z, Bai Y, Wan Ishak WZ, Shim BY, Park YL, Koo DH, Lu J, Xu J, Chon HJ, Bai LY, Zeng S, Yuan Y, Chen YY, Gu K, Zhong WY, Kuang S, Shih CS, Qin SK. Pembrolizumab versus paclitaxel for previously treated advanced gastric or gastroesophageal junction cancer (KEYNOTE-063): A randomized, open-label, phase 3 trial in Asian patients. Cancer. 2022 Mar 1;128(5):995-1003. doi: 10.1002/cncr.34019. Epub 2021 Dec 8. PMID 34878659
- See also: Merck Oncology Clinical Trial Information — http://keynoteclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2
Started | 47 | 47
Treated | 47 | 44
Completed | 0 | 0
Not Completed | 47 | 47
Not completed — Death | 44 | 46
Not completed — Study terminated by Sponsor | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2 | Total
Number analyzed (Participants) | 47 | 47 | 94
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.0 (10.4) | 59.0 (11.2) | 58.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 32 | 37 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 47 | 47 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 47 | 47 | 94
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Time to progression on first-line therapy [Count of Participants; unit: Participants]
  < 6 months | 30 | 30 | 60
  >= 6 months | 17 | 17 | 34
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS is graded on a scale from 0 (best) to 5 (worst). 0= fully active, able to carry on all pre-disease performance without restriction; 1= restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; 2= ambulatory and capable of all selfcare but unable to carry out any work activities (up and about more than 50% of waking hours); 3= capable of only limited selfcare; confined to bed or chair more than 50% of waking hours; 4= completely disabled, cannot carry on any selfcare, totally confined to bed or chair; 5= dead.
  Participants
    ECOG = 0 | 14 | 12 | 26
    ECOG = 1 | 33 | 35 | 68

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up.
Time Frame: Up to approximately 50 months
Population: Analysis population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 47 | 47
Months | 8.4 [4.0 to 9.5] | 7.7 [5.4 to 11.3]
Statistical Analysis 1: Comparison: Pembrolizumab 200 mg vs Paclitaxel 80 mg/m^2; Test type: Superiority; p = 0.2900, Log Rank; One-sided p-value based on log-rank test stratified by time to progression on first line therapy (< 6 months vs. ≥ 6 months) and ECOG PS (0 vs. 1); Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.58 to 1.36] — Based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by time to progression on first line therapy (< 6 months vs. ≥ 6 months) and ECOG PS (0 vs. 1)

2. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first. Per RECIST 1.1, progressive disease was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: The appearance of one or more new lesions was also considered progression. PFS as assessed by blinded independent central review will be presented.
Time Frame: Up to approximately 50 months
Population: Analysis population includes all randomized participants.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 47 | 47
Months | 1.9 [1.4 to 2.8] | 4.0 [2.7 to 6.2]
Statistical Analysis 1: Comparison: Pembrolizumab 200 mg vs Paclitaxel 80 mg/m^2; Test type: Superiority; p = 0.9954, Log Rank; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.77, 95% CI 2-sided [1.14 to 2.74] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per RECIST 1.1
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters) per RECIST 1.1.
Time Frame: Up to approximately 50 months
Population: Analysis population includes all randomized participants.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 47 | 47
Percentage of participants | 12.8 [4.8 to 25.7] | 19.1 [9.1 to 33.3]
Statistical Analysis 1: Comparison: Pembrolizumab 200 mg vs Paclitaxel 80 mg/m^2; Test type: Superiority; p = 0.7884, Z-test; One-sided p-value for testing. H0: difference in % = 0 versus H1: difference in % > 0; Difference in percentage = -6.0, 95% CI 2-sided [-21.6 to 9.3] — Based on Miettinen & Nurminen method stratified by time to progression on first line therapy (< 6 months vs. ≥ 6 months) and ECOG PS (0 vs. 1)

4. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An adverse event is defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to approximately 50 months
Population: Analysis population includes all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 47 | 44
Participants | 46 | 43

5. Secondary Outcome: Number of Participants Who Discontinue Study Treatment Due to an AE
Description: as for outcome 4
Time Frame: Up to approximately 25 months
Population: Analysis population includes all randomized participants who received at least one dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 47 | 44
Participants | 2 | 7

ADVERSE EVENTS:
Time Frame: Up to approximately 50 months
Description: All-cause mortality includes all randomized participants; Adverse events tables include all participants who received at least one dose of study drug. Per protocol, MedDRA preferred terms "Neoplasm Progression", "Malignant Neoplasm Progression" and "Disease Progression" not related to the drug are excluded.
Arm/Group | Pembrolizumab 200 mg | Paclitaxel 80 mg/m^2
All-Cause Mortality (participants affected / at risk) | 44/47 | 46/47
Serious Adverse Events (participants affected / at risk) | 13/47 | 14/44
Other Adverse Events (participants affected / at risk) | 46/47 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=47) | Paclitaxel 80 mg/m^2 (N=44)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 3 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 3 (3)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Thyroiditis (Endocrine disorders) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab 200 mg (N=47) | Paclitaxel 80 mg/m^2 (N=44)
Anaemia (Blood and lymphatic system disorders) | 17 (21) | 20 (26)
Granulocytopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (17)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 4 (22)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 6 (19)
Hyperthyroidism (Endocrine disorders) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 5 (5) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 4 (5) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 11 (12) | 6 (9)
Abdominal pain upper (Gastrointestinal disorders) | 6 (7) | 7 (8)
Ascites (Gastrointestinal disorders) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 7 (8) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 8 (21) | 8 (8)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (11) | 9 (10)
Vomiting (Gastrointestinal disorders) | 8 (11) | 4 (7)
Asthenia (General disorders) | 6 (7) | 6 (6)
Fatigue (General disorders) | 9 (9) | 7 (9)
Influenza like illness (General disorders) | 1 (1) | 3 (3)
Oedema peripheral (General disorders) | 4 (4) | 3 (4)
Pyrexia (General disorders) | 8 (9) | 7 (11)
Pneumonia (Infections and infestations) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (6)
Alanine aminotransferase increased (Investigations) | 5 (5) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 7 (7)
Blood albumin decreased (Investigations) | 3 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 9 (10) | 1 (1)
Blood bilirubin increased (Investigations) | 4 (5) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 7 (7) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 17 (55)
Weight decreased (Investigations) | 5 (5) | 4 (4)
White blood cell count decreased (Investigations) | 1 (1) | 13 (49)
Decreased appetite (Metabolism and nutrition disorders) | 5 (5) | 16 (19)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 14 (16) | 6 (7)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 3 (6)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Hypoproteinaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 4 (5)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 21 (21)
Pruritus (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (2):
  • Study Protocol (2020-04-22): https://cdn.clinicaltrials.gov/large-docs/88/NCT03019588/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT03019588/SAP_001.pdf